CLINICAL TRIAL: NCT05715970
Title: ICT Tools for the Diagnosis of Autoimmune Diseases in the Mediterranean Area_CAPITALISATION PROJECT
Brief Title: ICT Tools for the Diagnosis of Autoimmune Diseases
Acronym: ITAMA_CAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, Associate Professor, University of Palermo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ACPM32
Record Dates: First submitted 2023-01-18; First posted 2023-02-08 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; Point-of-Care-Test; Diagnosis
MeSH Terms: conditions — Celiac Disease; Disease

STUDY DESIGN:
Intervention Model Description: The ITAMA_CAP project, designed as a prospective, multicenter study [U.O.C. of Geriatrics (21.01) of the University Hospital of Palermo and the "Mater Dei" Hospital of Malta), provides for the enrollment of about 25,000 subjects, divided between Sicily and Malta. Approximately 10,000 students aged between 12 and 18 will be enrolled in Malta and approximately 15,000 adults (>18 years) will be enrolled in Sicily. These numbers are dictated by the need to obtain heterogeneous samples comparable with the subjects diagnosed in the previous ITAMA project (20,000). In Sicily, screening will be carried out in the GPs (Italian takers) clinics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- General population (Experimental): 25,000 subjects, divided between Sicily and Malta. Approximately 10,000 students aged between 12 and 18 will be enrolled in Malta and approximately 15,000 adults (>18 years) will be enrolled in Sicily. These numbers are dictated by the need to obtain heterogeneous samples comparable with the subjects diagnosed in the previous ITAMA project (20,000). In Sicily, screening will be carried out in the GPs (Italian takers) clinics. In Malta the recruitment will be performed in the schools (Maltese takers). Furthermore, in Malta, a further extension of the results provides for the execution of the PoCT+questionnaire in the asymptomatic first-degree relatives of the pediatric subjects with an ascertained diagnosis of CD identified in the previous project.
  Interventions: Diagnostic Test: PoCT+questionnaire administration

INTERVENTIONS:
Diagnostic Test: PoCT+questionnaire administration — In Sicily, screening will be carried out in the general practitioner's clinics (GPs). GPs will have to submit the patients attending their clinics to the PoCT + software tools questionnaire. Subjects who are PoCT positive and/or who reach the minimum score in the questionnaire will be considered 'patients at risk of CD' and must be subjected, with prior consent, to in-depth diagnostics using standard serological methods. The subjects resulting positive in the serological investigations will then undergo the appropriate endoscopic and biopsy investigations to ascertain the presence of CD. In Malta the recruitment will exactly repeat the modalities already carried out in the ITAMA project, through the schools of Malta (Maltese takers), while the laboratory and endoscopic examinations of the subjects who tested positive for the PoCT and/or who will reach the minimum score in the software tools questionnaire will be centralized at the "Mater Dei" hospital.

SUMMARY:
The ITAMA project, which ended in 03/2022, came from the need to increase/anticipate the number of diagnosed cases of celiac disease (CD). The project involved the preliminary development of 'software tools' (Graphical User Interface (GUI), DATABASE, Decision Support System (DSS)) used to support the physicians to optimize CD diagnosis. Subsequently, through a screening of about 20,000 subjects of school age in Malta and about 1,000 subjects in Sicily, it was shown that, in compliance with international guidelines, it is possible to anticipate CD diagnosis and make it easy with the aid of a tool based on the search for specific antibodies in the blood, collecting a single drop of blood - with a test performed directly "in the points where care is provided" (eg schools, outpatient clinics) that is with a Point-of-Care-Test (PoCT). This system proved to be effective, and the method was minimally invasive (at least in some pediatric cases it was possible to avoid the endoscopic examination).

The ITAMA project has made it possible to bring out a submerged part of the "CD iceberg", a condition that in a large percentage of cases remains undiagnosed and transfer the know-how to commercial companies in the medical sector.

ITAMA project results allowed to verify and validate, on a large sample of subjects subjected to screening, that:

1. Diagnosis can be anticipated and facilitated by combined use of a rapid test (PoCT), medical history (supported by software) and traditional serological tests.
2. The diagnosis can be optimized by the support of Information Technology (IT) tools based on Artificial Intelligence (AI).
3. Non-invasive methods, if correctly applied, allow CD diagnosis avoiding invasive diagnostic techniques.
4. The reported procedures grant considerable savings for the National Health System (NHS).

Starting from the results of ITAMA, this capitalization project aims to extend the previous experience in a larger population with heterogeneous characteristics (both adults and children).

The goal of the new project is to use the combination of PoCT + tools software, to increase/anticipate CD diagnosis and, therefore, bring the number of diagnosed subjects closer to the number of expected cases, in Sicily and Malta. The inevitable implication of this would be the improvement in the quality of life of patients (reduction of symptoms, fewer medical visits and instrumental examinations performed, reduction of lost working days, improvement of social relations) and a significant reduction in costs for the NHS.

DETAILED DESCRIPTION:
Background The diagnosis of celiac disease (CD), a known autoimmune disease, presupposes the recognition of symptoms/signs, the carrying out of serological tests and the diagnostic confirmation with histological examination of intestinal biopsies. The pediatric guidelines European Society for Pediatric Gastroenterology Hepatology and Nutrition report the possibility of avoiding biopsy in some classes of pediatric patients. It is estimated that about 1% of the world population is affected by CD, but only 0.37% of the Italian population and 0.40% in Malta, to date, has been diagnosed. In Sicily in particular, the cases not yet diagnosed are probably even more than in the rest of the Italian territory, because the prevalence was slightly lower than the national average (0.35%). It is clear from these data that CD is an underestimated pathology throughout the national territory and even more in Sicily. It is also known that CD is associated with various pathologies with an autoimmune component (including type 1 diabetes mellitus and Hashimoto's thyroiditis) and that, among its complications, more present in subjects who do not practice or are refractory to a gluten-free diet, neoplastic diseases are also included, such as intestinal T-cell lymphoma and small intestine adenocarcinoma.

The ITAMA project, which ended in March 2022, was born from the need to increase/anticipate the number of diagnosed cases of CD by optimizing its diagnosis. The project has developed 'software tools' (Graphical User Interface (GUI), DATABASE, Decision Support System (DSS)) to support the physicians in optimizing CD diagnosis. Through a screening, conducted on 20,000 school-age subjects in Malta and about 1,000 subjects in Sicily, it was demonstrated that, in compliance with the European Society Paediatric Gastroenterology, Hepatology and Nutrition guidelines, it was possible to anticipate the diagnosis of CD and make it easy with the aid of a test performed directly "at the points where treatment is provided" (e.g. schools, medical clinics), i.e. with a Point-of-Care-Test (PoCT, Celiac Disease Quick TestBIOHIT HealthCare Srl, Milan, Italy), conducted on capillary blood obtained through simple and low cost finger prick. This system has proved to be an effective, and the method to be minimally invasive and inexpensive making it possible, at least in certain pediatric cases, to bring out a submerged part of the "CD iceberg", avoiding further investigations, even invasive, in patients with negative PoCT. With ITAMA it was therefore possible to transfer the "know-how" to commercial companies in the medical sector, activating a network between research and production areas in the healthcare sector through the development of information and communication technologies (ICT) for the diagnosis of the CD. The results made it possible to verify/validate, on a large sample of subjects, that:

* the diagnosis can be anticipated/facilitated through the combined use of a rapid test (PoCT), medical history and traditional serological tests
* the diagnosis can be optimized thanks to the support of computer tools based on artificial intelligence (AI).

The capitalization of the aforementioned results is probably possible through the National Health System (NHS) and schools and could be strategic because:

* non-invasive methods, if correctly applied, allow an early and effective diagnosis of CD (currently underdiagnosed) and, in some cases, can also allow patients not to be subjected to invasive diagnostic methods
* the aforementioned procedures allow a considerable saving for the NHS.

Objectives The present project aims to capitalize and extend the previous experience of ITAMA in a larger population with heterogeneous characteristics (young people and adults), through the Sicilian network of General Practitioners (GPs) and the involvement of numerous schools in Malta .

The goal is to use ITAMA outputs/results to increase/anticipate the diagnosis of CD and, therefore, bring the number of diagnosed subjects closer to the expected number of CD cases in Sicily and Malta. The consequence could be the improvement of the quality of life of the diagnosed patients (anticipation of diagnosis and therapy, with consequent reduction of symptoms/signs, reduction of medical visits/instrumental tests performed, reduction of lost working days, improvement of social relationships) and a significant reduction in costs for the NHS, as well as a reduction in the number of conventional tests (laboratory and instrumental investigations) not recommended in patients with negative PoCT and the further consequent costs caused by these.

Expected results The expected results from this "extension" of the ITAMA project would essentially consist in the capitalization of the previously observed results, through: A) the involvement of the Sicilian network of GPs and Maltese schools and their greater knowledge and awareness of the need to bring out the diagnoses miss you today; B) the confirmation of a possible and extensive outpatient use of the PoCT method to facilitate diagnosis.

From a clinical point of view, we also expect: 1) an increase in CD diagnoses, bridging the gap between diagnosed cases and estimated cases, also showing any differences in prevalence between adults and children; 2) a reduction in diagnostic delays, with a consequent improvement in the quality of life of patients and a reduction in costs for the NHS; 3) a reduction in the number of conventional tests (laboratory and instrumental investigations) not recommended in patients with negative PoCT and in the further consequent costs caused by these.

From a scientific point of view, this study will contribute to: 1) define more precisely the prevalence of CD in two populations of the Mediterranean area; 2) create a database usable by researchers for this and future research; 3) to demonstrate the utility of a minimally invasive and low-cost screening test for the early identification of patients with CD.

ELIGIBILITY:
Inclusion Criteria:

* age >12 and <18 years for subjects enrolled in Malta;
* age >18 years for subjects enrolled in Sicily.

Exclusion Criteria:

* age <12 and >18 years for subjects enrolled in Malta;
* age <18 years for subjects enrolled in Sicily;
* refusal to undergo the proposed diagnostic procedures;
* lack of informed consent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25000 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of subjects testing positive to PoCT. | 1 day
  Point-of-Care-Test (PoCt) will be performed on all subjects recruited at General Practitioner's clinics in Sicily and at schools in Malta. Whole blood sample will be collected by puncture of the index, middle or ring finger. The blood must be dispensed slowly onto the test cassette, where there is a special oval indicated by an arrow. After 30-60 seconds two drops of buffer diluent should be added in the same window. After 10 minutes, the healthcare professional will be able to read the test. Reading Test Results: NEGATIVE: Only one BLUE band appears in the Results Window near the letter "C" (control line) of the Test Cassette. This band must always appear. POSITIVE: In addition to the BLUE control band, a discernible PINK-RED band also appears in the result window near the letter "T" (test line) of the test cassette. The intensity of the line depends on the concentration of antibodies in the blood. INVALID: absence of BLUE band in the results window near the letter "C".
Identification of subjects with probable CD by the use of software tools | 1 day
  A structured questionnaire to Celiac Disease (CD) symptoms, signs and predisposing factors (eg. familiarity, etc.) will be administered to all subjects recruited at General Practitioner's clinics in Sicily and at schools in Malta, by the use of the software tools developed in the ITAMA project. In particular, data entry into the Database, already implemented in the ITAMA project, can be managed through a GUI created in the Java language for greater product portability. The GUI allows the presentation of the outputs in a structured way and has, among its functions: a) the data acquisition mode (DAQ), b) the data search and consultation mode (QUERY) and c) the execution of the Decision Support System (DSS) for the diagnosis of CD.
  The DSS will provide an output according to the software elaboration as: 'Probable CD: further diagnostic testing is suggested' or 'Unlikely CD: no further diagnostic testing is suggested'.
Identification of patients positive to CD serological markers (IgA anti-tTg) | 2 weeks
  All patients who tested positive to PoCT and/or who had the 'Probable Celiac Disease: further diagnostic testing is suggested' output after the software tools elaboration will be subjected to the search for specific antibodies for celiac disease.
  Immunoglobulin A class anti-transglutaminase will be analyzed by commercial kits, on blood samples collected by venipuncture.
Identification of patients positive to CD serological markers (IgG anti-tTg) | 2 weeks
  All patients who tested positive to PoCT and/or who had the 'Probable Celiac Disease: further diagnostic testing is suggested' output after the software tools elaboration will be subjected to the search for specific antibodies for celiac disease.
  Immunoglobulin G class anti-transglutaminase will be analyzed by commercial kits, on blood samples collected by venipuncture.
Identification of patients positive to CD serological markers (EmA) | 2 weeks
  All patients who tested positive to PoCT and/or who had the 'Probable Celiac Disease: further diagnostic testing is suggested' output after the software tools elaboration will be subjected to the search for specific antibodies for celiac disease.
  Anti-Endomysial Antibody will be analyzed by commercial kits, on blood samples collected by venipuncture.
Identification of patients positive to CD histology | 4 weeks
  All patients who had serological tests compatible with Celiac Disease (immunoglobulin (Ig)A class anti-transglutaminase (tTg) and Anti-Endomysial Antibody (EmA) positivity in IgA-sufficient patients or IgG class anti-tTG and EmA in IgA-deficient subjects) will be subjected to esophago-gastro duodenoscopy and will be diagnosed as suffering from Celiac Disease according the results of histology examination (Marsh-Oberhuber classification).

CONTACTS AND LOCATIONS:
Locations (2):
- University Hospital of Palermo, Palermo, Sicily, Italy
- Mater Dei Hospital, Valletta, Malta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fasano A, Berti I, Gerarduzzi T, Not T, Colletti RB, Drago S, Elitsur Y, Green PH, Guandalini S, Hill ID, Pietzak M, Ventura A, Thorpe M, Kryszak D, Fornaroli F, Wasserman SS, Murray JA, Horvath K. Prevalence of celiac disease in at-risk and not-at-risk groups in the United States: a large multicenter study. Arch Intern Med. 2003 Feb 10;163(3):286-92. doi: 10.1001/archinte.163.3.286. PMID 12578508
- [Background] Mansueto P, Spagnuolo G, Calderone S, D'Agate CC, Cosenza S, Leonardi G, Camilleri S, Pistone M, Seminara G, Alaimo C, Soresi M, Carroccio A, Garufi S. Improving the diagnostic approach to celiac disease: Experience from a regional network. Dig Liver Dis. 2022 Jun;54(6):771-775. doi: 10.1016/j.dld.2021.11.016. Epub 2021 Dec 21. PMID 34952810
- [Background] Husby S, Koletzko S, Korponay-Szabo I, Kurppa K, Mearin ML, Ribes-Koninckx C, Shamir R, Troncone R, Auricchio R, Castillejo G, Christensen R, Dolinsek J, Gillett P, Hrobjartsson A, Koltai T, Maki M, Nielsen SM, Popp A, Stordal K, Werkstetter K, Wessels M. European Society Paediatric Gastroenterology, Hepatology and Nutrition Guidelines for Diagnosing Coeliac Disease 2020. J Pediatr Gastroenterol Nutr. 2020 Jan;70(1):141-156. doi: 10.1097/MPG.0000000000002497. PMID 31568151
- [Background] Magazzu G, Aquilina S, Barbara C, Bondin R, Brusca I, Bugeja J, Camilleri M, Cascio D, Costa S, Cuzzupe C, Duca A, Fregapane M, Gentile V, Giuliano A, Grifo A, Grima AM, Ieni A, Li Calzi G, Maisano F, Melita G, Pallio S, Panasiti I, Pellegrino S, Romano C, Sorce S, Tabacchi ME, Taormina V, Tegolo D, Tortora A, Valenti C, Vella C, Raso G. Recognizing the Emergent and Submerged Iceberg of the Celiac Disease: ITAMA Project-Global Strategy Protocol. Pediatr Rep. 2022 Jun 10;14(2):293-311. doi: 10.3390/pediatric14020037. PMID 35736659
- [Background] Catassi C, Fasano A. Celiac disease diagnosis: simple rules are better than complicated algorithms. Am J Med. 2010 Aug;123(8):691-3. doi: 10.1016/j.amjmed.2010.02.019. PMID 20670718
- [Background] Caio G, Volta U, Sapone A, Leffler DA, De Giorgio R, Catassi C, Fasano A. Celiac disease: a comprehensive current review. BMC Med. 2019 Jul 23;17(1):142. doi: 10.1186/s12916-019-1380-z. PMID 31331324